CLINICAL TRIAL: NCT01424943
Title: The Family Networks Project Study One: Supporting Family Confidence, Competence, and Community Connections
Brief Title: Family Networks Project Study One: An Efficacy Study of Stepping Stones Triple P for Children Under Age Two
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Quality Improvement Center for Early Childhood (Unknown)
Responsible Party: Principal Investigator, Cheri Shapiro, Ph.D., Research Associate Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00006462
Record Dates: First submitted 2011-07-27; First posted 2011-08-29 (Estimated); Results first posted 2014-12-15 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Prevent Child Maltreatment
Keywords: prevention; evidence-based parenting intervention; children; disabilities; IDEA Part C; Stepping Stones Triple P

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stepping Stones Triple P (Experimental): 10-15 sessions of Level 4 Standard Stepping Stones Triple P delivered in family homes
  Interventions: Behavioral: Stepping Stones Triple P
- BabyNet Services As usual (Other): BabyNet services as usual based on IFSP
  Interventions: Behavioral: Stepping Stones Triple P; Other: BabyNet Services As usual

INTERVENTIONS:
Behavioral: Stepping Stones Triple P — 10-12 session manualized intervention delivered in client homes
Other: BabyNet Services As usual — BabyNet services as usual based on IFSP
  Arms: BabyNet Services As usual

SUMMARY:
The purpose of the project is to assess the initial efficacy of Stepping Stones Triple P-Positive Parenting Program (SSTP) with parents of children below age two with developmental disabilities to strengthen families and prevent child maltreatment.

DETAILED DESCRIPTION:
This study is an initial efficacy trial of SSTP for parents of children below age 2. The target population consists of 50 families of young children ages 11-23 months with developmental disabilities who are eligible to receive IDEA Part C (Individuals with Disabilities Education Act Part C) services in one region of South Carolina. Families will be randomly assigned to one of two conditions (1) IDEA Part C services as usual or (2) IDEA Part C services plus SSTP. Project goals are to strengthen parent competence, enhance parent confidence, and strengthen child social, emotional and behavioral functioning. Ultimately, this should result in a reduced likelihood of child maltreatment

ELIGIBILITY:
Inclusion Criteria:

* child age between 11 and 23 months of age
* child eligible for IDEA Part C Services
* parent english speaking
* parent willing to allow in-home services

Exclusion Criteria:

* disability requiring extensive out of home treatment

Ages: 11 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2010-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cheri Shapiro, Ph.D., Principal Investigator — Research Associate Professor, Parenting and Family Research Center, University of South Carolina
Locations (1):
- Parenting and Family Research Center, Columbia, South Carolina, United States

REFERENCES:
- See also: Quality Improvement Center for Early Childhood — http://www.qic-ec.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Stepping Stones Triple P Plus IDEA Part C Services as Usual: 10-15 sessions of Level 4 Standard Stepping Stones Triple P delivered in family homes
  Stepping Stones Triple P: 10-12 session manualized intervention delivered in client homes. Families also recieved IDEA Part C early intervention services as usual per the family IFSP.
- IDEA Part C Services As Usual: IDEA Part C services as usual based on IFSP
Period: Overall Study
Arm/Group | Stepping Stones Triple P Plus IDEA Part C Services as Usual | IDEA Part C Services As Usual
Started | 25 | 24
Completed | 12 | 23
Not Completed | 13 | 1

BASELINE CHARACTERISTICS:
Population: Parents of children with disabilities eligible for IDEA Part C Services and their identified child
Groups:
- Total: Total of all reporting groups
Arm/Group | Stepping Stones Triple P Plus IDEA Part C Services as Usual | IDEA Part C Services As Usual | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Continuous [Mean (Standard Deviation); unit: months] | 18.77 (3.64) | 19.25 (3.13) | 19.00 (3.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 17 | 14 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 7 | 5 | 12
  White | 14 | 11 | 25
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 25 | 24 | 49

OUTCOME MEASURES:

1. Primary Outcome: Parenting Style
Description: Parenting Scale (Total Score; measure of parenting style). 30 items on the scale, scores range from 1-7 for each item with higher scores indicating dysfunctional parenting styles (laxness, over-reactivity, hostility). Scores summed and divided by 30 for total score.
Time Frame: Baseline, 5 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Stepping Stones Triple P Plus IDEA Part C Services as Usual | IDEA Part C Services As Usual
Number analyzed (Participants) | 25 | 24
scores on a scale
  baseline Parenting Scale | 2.65 (.57) | 2.61 (.70)
  Post-Tx Parenting Scale | 2.09 (.73) | 2.21 (.66)

2. Primary Outcome: Child Behavior
Description: Child Behavior Checklist 1/5-5. A parent report measure of child behavioral problems. The score used for this outcome was the CBCL Total Score, which is a T-Score. T scores average 50 with a standard deviation of 10. Scores above 65 considered in the clinical range.
Time Frame: Baseline, 5 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Stepping Stones Triple P Plus IDEA Part C Services as Usual | IDEA Part C Services As Usual
Number analyzed (Participants) | 25 | 24
T-score
  CBCL Total Score Baseline | 53.56 (8.54) | 51.00 (10.67)
  CBCL Total Score Post-Tx | 53.45 (10.91) | 51.61 (9.09)

3. Primary Outcome: Parenting Self-confidence
Description: Toddler Care Questionnaire. Measures parent reported self-confidence in parenting a toddler. Parents rate their confidence in performing parenting tasks specific to toddlers. Higher scores indicate more confidence. Scores range from 37-185. The total sum score derived from adding the scores for the 37 items in this survey was used for this outcome measure.
Time Frame: Baseline, 5 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stepping Stones Triple P Plus IDEA Part C Services as Usual | IDEA Part C Services As Usual
Number analyzed (Participants) | 25 | 24
units on a scale
  baseline | 152.32 (21.93) | 155.13 (19.19)
  midpoint | 157.45 (19.68) | 159.17 (14.65)

4. Primary Outcome: KIPS
Description: KIPS observational measure of the quality of the parent-child relationship. scores range from 1-5. Higher scores indicate a higher quality of relationship.
Time Frame: Baseline, 5 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Stepping Stones Triple P Plus IDEA Part C Services as Usual | IDEA Part C Services As Usual
Number analyzed (Participants) | 25 | 24
scores on a scale
  Scores at 5 months | 3.52 (.70) | 3.52 (.63)
  scores at Baseline | 3.39 (.54) | 3.52 (.59)

5. Secondary Outcome: Parent Symptoms of Depression, Anxiety and Stress
Description: DASS-21, brief screening measure of symptoms of depression, anxiety, and stress. Scores on each scale range from 0-21. Higher scores indicate more symptoms in each area.
Time Frame: baseline, 5 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Stepping Stones Triple P Plus IDEA Part C Services as Usual | IDEA Part C Services As Usual
Number analyzed (Participants) | 25 | 24
scores on a scale
  5 month DASS 21 Depression | 3.00 (4.22) | 4.09 (5.92)
  5 month DASS 21 Anxiety | 3.45 (3.56) | 2.96 (5.25)
  5 month DASS 21 Stress | 9.55 (6.35) | 10.70 (9.12)
  baseline DASS 21 depression | 4.80 (6.16) | 4.58 (9.16)
  baseline DASS 21 anxiety | 3.68 (5.59) | 3.50 (7.11)
  baseline DASS 21 stress | 11.20 (6.98) | 10.83 (8.50)

ADVERSE EVENTS:
Arm/Group | Stepping Stones Triple P Plus IDEA Part C Services as Usual | IDEA Part C Services As Usual
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 0/25 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No